CLINICAL TRIAL: NCT02872584
Title: Serum Free Fatty Acids Desaturase Activity Indices in Sera of Patients on Long-term High-dose Corticosteroid Treatment
Brief Title: Serum FFA Desaturase Activity Index in Patients on High Dose Corticosteroids
Acronym: FFA&steroids
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Irit HOCHBERG MD, Attending Physican, Institute of Diabete Endocrinology and Metabolism, Rambam Health Care Campus
Other Study IDs: 0134-16-RMB CTIL
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Glucocorticoid
MeSH Terms: interventions — Prednisone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prednisone: Patients with dermatological conditions requiring high dose long term glucocorticoid treatment
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Prednisone — prednisone treatment as required by dermatological condition (pemphigus/pemphigoid)

SUMMARY:
Free fatty acid index will be measured in patients before and 1 month after high dose prednisone.

DETAILED DESCRIPTION:
Serum Free Fatty Acids Desaturase Activity Indices in Sera of Patients with Pemphigus and Bullous Pemphigoid on Long-term High-dose Corticosteroid Treatment

1.1 BACKGOUND & STUDY RATIONALE Chronic exposure to glucocorticoids exerts profound effects on subcutaneous and visceral adipose tissues, and may induce both lipolysis and lipogenesis [1].

In acute conditions (such as stress) glucocorticoids increase whole body lipolysis, and free fatty acid production and turnover. However, in chronic glucocorticoid excess conditions (such as Cushing's syndrome), this acute induction of systemic lipolysis is not sustained, and actually decreases. Moreover, glucocorticoids may act synergistically with insulin to upregulate lipogenesis, and increase triglycerides storage, mainly in the liver and visceral adipose tissue [2, 3]

Increased subcutaneous fat mass is a hallmark of Cushing's syndrome and could potentially be mediated through the activation of lipogenesis. We have recently published a study that found an upregulation of free fatty acids synthesis and desaturases genes and triglyceride synthesis genes in subcutaneous adipose tissue from subjects with Cushing's disease, further supporting the hypothesis that lipogenesis is activated in these tissues via the transcriptional activation of fatty acid synthesis and triglyceride synthesis [4]. In parallel, we saw higher levels of lipolysis in adipose tissue explants from Cushing's disease patients [4].

In general, serum free fatty acids composition is influenced by dietary fat intake, desaturating enzymes activity (in subcutaneous and visceral adipose tissues, and liver), insulin resistance and lifestyle factors such as physical activity, and obesity [5, 6, 7]. However, fasting serum free fatty acids are not directly derived from nutritional intake, but primarily originate from adipose tissue storages [8, 9] Desaturase indices, estimated as product-to-precursor fatty acid ratios, are employed in epidemiological studies. Desaturase activity indices were estimated according to the following: Stearoyl-CoA desaturase-16 (SCD-16) = 16:1(n-7) / 16:0, Stearoyl-CoA-desaturase-18 (SCD-18) = 18:1(n-9) / 18:0, Delta-5-desaturase (D6D) = 20:3(n-6) / 18:2 (n-6), and Delta-5-desaturase (D5D) = 20:4(n-6) / 20:3 (n-6).

Estimated SCD-16, SCD-18, and D5D activity ratios were found to be correlated between fasting serum free fatty acids and subcutaneous adipose tissue triglycerides [10]. Moreover, the subcutaneous adipose tissue estimated SCD-16, and SCD-18 activity ratios, were significantly correlated with SCD gene expression in this tissue [11].

Long-term effects of glucocorticoids on serum fasting free fatty acids composition and desaturase indices were not studied. Our goal in this study is to examine whether there are significant changes in estimated serum free fatty acids desaturase indices and in total free fatty acids and glycerol after long-term glucocorticoid therapy.

1.2 STUDY OBJECTIVES 1.2.1 Primary objective The primary objective of this study is to compare desaturase activity indices in sera of patients with pemphigus and bullous pemphigoid, collected before, and one month after the initiation of high-dose oral corticosteroid treatment.

Secondary objectives The secondary objectives are to examine the changes in weight, waist/hip ratio, insulin resistance as reflected by the HOMA-IR model, and fasting lipid profiles, over one month of high-dose oral corticosteroid treatment.

1.3 STUDY DESIGN This is a single-center prospective cohort study.

1.3.1 Study population About 20 consecutive eligible patients diagnosed with pemphigus or bullous pemphigoid, who are planned to be placed on a high dose oral corticosteroid regimen (equivalent to 0.5mg/kg/day or more of prednisone) for at least one month, will be recruited.

1.3.2 Study duration Total duration of the study is expected to be 10 months.

1.4 STUDY METHODS For each patient, blood samples will be collected before, and one month after the initiation of high-dose oral corticosteroids. Serum samples will be collected in the morning after overnight fasting of approximately 12 hours.

Each blood sample will be assessed for the following:

- Serum free fatty acids levels, including: Palmitoleic Acid (16:1(n-7)), Palmitic Acid (C16:0), Oleic Acid (C18:1(n-9)), Stearic Acid (C18:0), Linoleic Acid (C18:2(n-6)), Arachidonic Acid (C20:4(n-6)), and Dihomogamma Linolenic (C20:3(n-6)).

Free fatty acids Levels in serum will be determined using Gas Chromatography-Mass Spectrometry (GC/MS) Stable Isotope Dilution Analysis kit.

* Fasting lipid profile: Total cholesterol, low-density lipoprotein (LDL), high-density lipoprotein (HDL), Triglycerides (TG), and free glycerol.
* Fasting plasma glucose, plasma insulin, and glycated hemoglobin (HbA1c)
* Complete blood count
* Creatinine and Urea
* Albumin and total protein
* Liver enzymes: AST, ALT, GGT, ALP
* Thyroid hormones: TSH, FT4, FT3

Desaturase activity indices will be estimated according to the following:

* Stearoyl-CoA desaturase-16 (SCD-16) = 16:1(n-7) / 16:0
* Stearoyl-CoA-desaturase-18 (SCD-18) = 18:1(n-9) / 18:0
* Delta-5-desaturase (D6D) = 20:3(n-6) / 18:2 (n-6)
* Delta-5-desaturase (D5D) = 20:4(n-6) / 20:3 (n-6).

Insulin resistance will be estimated by HOMA-IR (fasting insulin (mU/l) × fasting glucose (mmol/l)/22.5).

The following physical measurements will be taken at enrolment and one month later:

* Weight, Height (BMI)
* Waist and hip measurement (waist/hip ratio)

ELIGIBILITY:
Inclusion Criteria:

* Each participant must be at least 18 years of age.
* Each participant must give a written informed consent for participation in the study.
* Each participant must be drug naïve with respect to previous glucocorticoid treatment (history of less than 2-week treatment at any time is authorized, but with no recent glucocorticoid therapy over 3 months before study entry).

Exclusion Criteria:

* Obese subjects, defined as BMI > 35 or underweight subjects, defined as BMI < 18.5
* A history of eating disorder
* Diabetes mellitus
* A history of Cushing's syndrome, subclinical hypercortisolism, hypoadrenalism, or congenital adrenal hyperplasia
* Abnormal thyroid function test : history of hyperthyroidism or hypothyroidism
* Active cancer
* Uncontrolled hypertension >160/95
* Hypercholesterolemia, defined as LDL > 190
* Hypertriglyceridemia, defined as TG > 250
* Acute or Chronic renal failure (GFR < 45) or nephrotic syndrome
* Acute or chronic hepatitis or cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: About 20 consecutive eligible patients diagnosed with pemphigus or bullous pemphigoid, who are planned to be placed on a high dose oral corticosteroid regimen (equivalent to 0.5mg/kg/day or more of prednisone) for at least one month, will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
free fatty acid quantification | 1 month

SECONDARY OUTCOMES:
insulin resistance | 1 month
weight gain | 1 month

IPD SHARING:
Plan to Share IPD: Yes